CLINICAL TRIAL: NCT05533164
Title: Rituximab Effect on Decreasing glUcoCorticoid Exposition in PolyMyalgia Rheumatica Patients Experiencing a PMR Relapse
Acronym: REDUCE-PMR-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Dutch Arthritis Association (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REDUCE-PMR-2
Record Dates: First submitted 2022-09-06; First posted 2022-09-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Polymyalgia Rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab (Experimental): 1000mg rituximab intravenously once
  Interventions: Drug: Rituximab
- Placebo (Placebo Comparator): 0mg rituximab (placebo) intravenously once
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rituximab — 1000mg rituximab in 250ml NaCl 0.9% intravenously
  Other Names: Rixathon; MabThera; Ruxience; Truxima
  Arms: Rituximab
Drug: Placebo — Placebo in 250ml NaCl 0.9% intravenously
  Arms: Placebo

SUMMARY:
Polymyalgia rheumatica (PMR) is prevalent among elderly. Untreated, it leads to major reduction in quality of life. Glucocorticoids are the cornerstone of treatment, but have drawbacks, warranting glucocorticoid sparing treatment. A proof of concept study on Rituximab (RTX) vs placebo showed efficacy in 48 vs 21%(p=0.049) in glucocorticoid free remission after 21 weeks (Marsman et al. 2021). Though promising, the short study duration, small sample size and only few relapsing patients included in this study require further confirmation. Therefore a larger randomised controlled trial with longer follow up will be performed on RTX efficacy on glucocorticoid free remission in relapsing PMR patients during glucocorticoid taper.

ELIGIBILITY:
Inclusion Criteria:

* Polymyalgia rheumatica (PMR) diagnosis fulfilling the 2012 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria
* Experiencing a PMR relapse, defined as recurring of symptoms and increase in erythrocyte sedimentation rate (ESR)/ C reactive protein (CRP)
* Unable to reduce glucocorticoid dose below 5mg/day prednisolone or equivalent
* Informed consent

Exclusion Criteria:

* Treatment with systemic immunosuppressants (other than GC, MTX, leflunomide and azathioprine) 3 months prior to inclusion;
* (clinical) suspect concomitant giant cell arteritis or other rheumatic inflammatory diseases;
* concomitant conditions that might significantly interfere with PMR pain or movement evaluation as judged by the investigator;
* previous hypersensitivity for RTX or contra-indications to RTX.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Between group difference in percentage of patients in glucocorticoid-free remission | At week 52
  Between group difference in percentage of patients in glucocorticoid-free remission (PMR activity score < 10) at week 52

SECONDARY OUTCOMES:
Percentage of patients in glucocorticoid-free remission | 21 weeks
  Percentage of patients in glucocorticoid-free remission
Percentage of patients with glucocorticoid dose of ≤5mg/day | 52 weeks
  Percentage of patients with glucocorticoid dose of ≤5mg/day
Number of relapses | 52 weeks
  Number of relapses
Time to glucocorticoid-free remission | 52 weeks
  Time to glucocorticoid-free remission in days during the study period
Time to relapse | 52 weeks
  Time to relapse in days during the study period
Cumulative glucocorticoid dose | 52 weeks
  Cumulative glucocorticoid dose
Percentage of patients needing RTX/Placebo retreatment | 52 weeks
  Percentage of patients needing RTX/Placebo retreatment
Adverse events | 52 weeks
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Aatke van der Maas, Principal Investigator — Sint Maartenskliniek
Locations (1):
- Sint Maartensklineik, Ubbergen, Gelderland, Netherlands

REFERENCES:
- [Derived] Sun MM, Pope JE. Polymyalgia rheumatica and giant cell arteritis: diagnosis and management. Curr Opin Rheumatol. 2025 Jan 1;37(1):32-38. doi: 10.1097/BOR.0000000000001059. Epub 2024 Oct 14. PMID 39400109